CLINICAL TRIAL: NCT01221454
Title: Efficacy of Allogenic Bone Marrow Stem Cells Transplantation in Patients With Liver Failure Resulting From Chronic Hepatitis B
Brief Title: Allogenic Bone Marrow Stem Cell Transplantation in Liver Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Lin Bingliang, Third Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS-LF
Record Dates: First submitted 2010-10-12; First posted 2010-10-15 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Liver Failure
Keywords: ABMSC; Allogenic bone marrow mesenchymal stem cells; Liver Failure; Transplantation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A(conserved therapy ) (Active Comparator): Thirty of the enrolled patients were assigned to Group A to receive comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine.
  Interventions: Drug: Conserved therapy
- Group B (BMSC Transplantion) (Experimental): Thirty of the enrolled patients were assigned to Group B to receive comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine, as well as bone marrow stem cells transplantation
  Interventions: Procedure: Allogenic bone marrow stem cells transplantation

INTERVENTIONS:
Procedure: Allogenic bone marrow stem cells transplantation — 30ml allogenic bone marrow stem cells were infused to patients using interventional method via portal vein or hepatic artery as well as conserved therapy
  Arms: Group B (BMSC Transplantion)
Drug: Conserved therapy — Oral or intravenous administration
  Arms: Group A(conserved therapy )

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy of allogenic bone marrow stem cells (BMSCs) transplantation in patients with liver failure caused by hepatitis B infection. The evaluation of the efficacy includes the level of serum alanine aminotransferase (ALT), aspartate aminotransferase(AST), total bilirubin (TB),prothrombin time (PT), albumin (ALB), prealbumin(PA), liver histological improvement before and 1 week to 1 year after transplantation. Child-Pugh scores, MELD scores and clinical symptoms were also observed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16~65 years.
* Serum HBsAg positive for over six months.
* Meet the diagnostic criteria of liver failure:

Exclusion Criteria:

* History of moderate to severe hepatic encephalopathy or variceal bleeding during the last two months before enrolment.
* Prothrombin time is over 30s.
* Cirrhosis caused by other reasons except HBV infection.
* Severe problems in other vital organs(e.g.the heart,renal or lungs).
* Liver tumor on ultrasonography, CT or MRI examination.
* Pregnant or lactating women.
* Imaging evidences of vascular thromboses.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Liver Function | 12 months
  The levels of serum alanine aminotransferase (ALT), total bilirubin (TB),prothrombin time (PT), albumin (ALB), prealbumin(PA), number of leucocyte,erythrocyte and platelet, cytokines, T lymphocyte and B lymphocyte,liver histological

SECONDARY OUTCOMES:
Immune function | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: The Third Affiliated Hospital of Sun Yat-sen University — http://www.zssy.com.cn/